CLINICAL TRIAL: NCT00651391
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Effect of Ezetimibe Plus Simvastatin Compared With Simvastatin Alone on Flow-Mediated Brachial Artery Vasoactivity in Subjects With Primary Hypercholesterolemia (The EFFECTS Trial)
Brief Title: Effect of Ezetimibe Plus Simvastatin on Flow-Mediated Brachial Artery Vasoactivity in Subjects With Primary Hypercholesterolemia (Study P03336)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: P03336
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Atherosclerosis
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis | interventions — Ezetimibe, Simvastatin Drug Combination; Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ezetimibe + Simvastatin (Experimental)
  Interventions: Drug: Ezetimibe + Simvastatin
- Simvastatin (Active Comparator)
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ezetimibe + Simvastatin — oral tablet of ezetimibe 10 mg plus simvastatin 20 mg once daily in the evening for 12 weeks
  Other Names: SCH 58235
  Arms: Ezetimibe + Simvastatin
Drug: Simvastatin — oral simvastatin 20 mg once daily in the evening for 12 weeks
  Arms: Simvastatin
Drug: Placebo — oral placebo once daily in the evening for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of ezetimibe coadministered with simvastatin compared with simvastatin alone when administered for 12 weeks on endothelial function as assessed by brachial artery reactivity testing (BART) using high-frequency ultrasound to image the brachial artery vasomotor response to a flow-mediated stimulus (high-shear stress) in subjects with high cholesterol. The secondary objectives include evaluation of nitroglycerin-induced vasodilation. In addition, lipid parameters (low-density-lipoprotein cholesterol [LDL-C], high-density-lipoprotein cholesterol [HDL-C], triglycerides [TG], total cholesterol [TC]) and C reactive protein (CRP) will be assessed by treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years old and older) with primary hypercholesterolemia with a plasma LDL-C >=145 mg/dL and <=250 mg/dL, and plasma TG <=350 mg/dL after adequate drug washout.
* Postmenopausal women who are receiving postmenopausal hormonal therapy or raloxifene must be maintained on a stable hormone replacement therapy (HRT) or raloxifene regimen for at least 6 weeks prior to study entry and throughout the study period.
* All subjects must agree to refrain from drinking alcohol or caffeine containing beverages for 12 hours prior to each study visit at which a BART assessment is performed; be minimally active (eg, avoid excessive physical activity) for 12 hours prior to each study visit at which a BART assessment is performed; and be willing to observe the NCEP Step I diet, participate in the study, and complete all study-related procedures.

Exclusion Criteria:

* Pregnancy or any other situation, condition, or illness that, in the opinion of the investigator, may interfere with optimal participation in the study
* Smoking, excessive alcohol consumption, underlying disease likely to limit life span to less than one year, or known hypersensitivity or any contraindication to simvastatin, ezetimibe, or nitroglycerin
* Existing hypercholesterolemia for which withholding approved lipid-lowering therapy for the duration of the study would be inappropriate
* The following concomitant illnesses: congestive heart failure NYHA Class III or IV; obstructive cardiomyopathy; uncontrolled cardiac arrhythmias; severe aortic stenosis; upper severe aortic stenosis; MI, CABG, or angioplasty within 6 months of study entry; uncontrolled hypertension; unstable or severe peripheral artery disease within 3 months of study entry; unstable angina pectoris; disorders of the hematologic, digestive or central nervous systems including cerebrovascular disease and degenerative disease that would limit study evaluation or participation; uncontrolled or newly diagnosed (within one month of study entry) diabetes mellitus; uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins (clinically euthyroid subjects on stable replacement doses of thyroid hormone are eligible for enrollment); known impairment of renal function (plasma creatinine >2.0 mg/dL), dysproteinemia, nephrotic syndrome or other renal disease (24-hour urinary protein 3+ or 1 gram); hepatobiliary or hepatic disease (subjects with AST or ALT >2 times the upper limit of reference range will be excluded); HIV positive; and known coagulopathy.
* Use of certain drugs, foods, or other agents known to alter lipid levels or to cause interactions with either ezetimibe or simvastatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-10-01 (Actual); Primary Completion 2004-09-01 (Actual); Study Completion 2004-09-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint in flow-mediated vasodilation: percent change in the mean diameter between 1-minute, post-cuff release diameter and image obtained prior to cuff application. | Week 12

SECONDARY OUTCOMES:
Change from baseline to endpoint in NTG-induced vasodilation: percent change in the diameter between the post-NTG and pre-NTG diameters. | Week 12
Changes from baseline to endpoint in LDL-C, HDL-C, TG, TC, and CRP. | Week 12